CLINICAL TRIAL: NCT04513756
Title: A Randomized Controlled Trial (RCT) to Asses the Efficacy of Community Reinforcement Approach (CRA) in the Treatment of Cannabis Users
Brief Title: Efficacy of Community Reinforcement Approach (CRA) in the Treatment of Cannabis Users
Acronym: Lifecare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Islamic University, Islamabad (Other)
Collaborators: Pakistan Institute of Living and Learning (Other)
Responsible Party: Principal Investigator, Muhammad Tahir Khalily, Professor of Clinical Psychology, International Islamic University, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9048/Federal/NRPU/R&D/HEC/2017
Record Dates: First submitted 2020-08-09; First posted 2020-08-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment Group (Experimental): Community Reinforcement Approach (CRA) as an intervention consisting of nine sessions (each session consists of 45-minutes). Treatment is primarily based upon the guidelines by Robert Meyers and William Miller (2001). The techniques included in the sessions are functional analysis, sobriety sampling, behavioral skills, and relapse prevention techniques.
  Interventions: Behavioral: Community Reinforcement Approach
- Treatment As Usual Group (No Intervention): CRA comprising of nine sessions will not be provided to this group. However, patients who will be already receiving treatment from any psychiatric or some other rehabilitation facility will be advised to continue their routine treatment.

INTERVENTIONS:
Behavioral: Community Reinforcement Approach — Community Reinforcement Approach (CRA) as an intervention consisting of nine sessions (each session consists of 45-minutes). Treatment is primarily based upon the guidelines by Robert Meyers and William Miller (2001). The techniques included in the sessions are functional analysis, sobriety sampling, behavioral skills, and relapse prevention techniques. The first three sessions of the intervention are based upon rapport building, induction of the rationale of CRA and Functional analysis of usage and non-usage behavior.
  Arms: Active Treatment Group

SUMMARY:
Substance abuse is not a new phenomenon in Pakistan. Its prevalence is increasing day by day due to multi-factorial reasons including psychological, cultural, biological, environmental, social and personal factors. Recent statistics shows an alarming increase in the use of substance. The last survey conducted indicates there are 3.6 million substance users in Pakistan and 3.6 percent among them are cannabis users. Furthermore, cannabis is found to be the most prevalent abused drug with adverse impact on the mental health among university students in Pakistan. However, there is a dearth of literature which could indicate a well-established treatment policy with proven efficacy model available in Pakistan. This study aims to investigate the efficacy of Community Reinforcement Approach (CRA) as evidence based remedy for Cannabis Users. The study is designed in a Randomized Controlled Trial (RCT) consisting of groups: Active Treatment (AT; with nine sessions of CRA intervention) and Treatment as Usual (TAU; routine treatment). After screening and baseline, participants will be assigned to the either Active Treatment group or Treatment As Usual group. Participants in both groups will be assessed on completion of third month after randomization (Outcome assessment), six months after randomization (first follow-up), and finally ninth months after randomization (second follow up). The primary outcome measure will be the frequency of usage, abstinence period and quantity of cannabis by using Timeline Follow Back Interview. The duration of the study is two and half years

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-30.
2. Current, regular cannabis use, defined as the use of any cannabis product at least twice per week over the course of the past 12 months.
3. Participant able to provide informed consent and willing to participate in the study.

Exclusion Criteria:

1. ICD-11 dependence (in the previous 12 months) on alcohol or any other illicit drug (apart from cannabis) with symptoms of withdrawal, tolerance or craving.
2. Current use of opiate substitution or sedative-hypnotic medication.
3. Having been treated for cannabis use problems with any other treatment within the previous three months.
4. Participant with lifetime psychotic disorder.
5. Participants with moderate, severe and extremely severe scores on (DASS-21) will be excluded. Severe learning disability or a pervasive developmental disorder.
6. Signs of severe non-cannabis-related intoxication.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-18 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
Time Line Follow-Back Interview (Assessing Change) | Participants in both groups will be assessed on baseline, completion of third month after randomization (Outcome assessment), six months after randomization (first follow-up), and finally ninth months after randomization (second follow up).
  In order to gather additional information about the frequency, patterns, mode and quantity of cannabis use, we will use the Time Line Follow-Back Interview (TLFB; Sobell & Sobell, 1992) as modified by the Marijuana Treatment Project Research Group, 2004, at baseline, prior to each therapy session, at post-treatment as well as at the follow-up assessments.
The Severity of Dependence Scale (Assessing Change) | Participants in both groups will be assessed on baseline, completion of third month after randomization (Outcome assessment), six months after randomization (first follow-up), and finally ninth months after randomization (second follow up).
  The Severity of Dependence Scale (SDS; Gossop, Darke, Griffiths, Hando, Powis, Hall, & Strang, 1995) will used to measure the degree of physical dependence the cannabis users experienced as well as the psychological components of their dependence. The scale will be used both at the time of screening and follow-ups.

SECONDARY OUTCOMES:
Depression Stress and Anxiety Questionnaire | Participants in both groups will be assessed on baseline, completion of third month after randomization (Outcome assessment), six months after randomization (first follow-up), and finally ninth months after randomization (second follow up).
  Depression Stress and Anxiety Questionnaire (Lovibond & Lovibond, 1995) will be used to measure depression, anxiety and stress in the participants. It is 21 item scales with 4 point rating (0-3). This scale will be used at the time of screening and follow-ups. Participants score falling in the category of severe to extremely severe will be excluded from the research at the time of screening.
EQ-5D-5L | Participants in both groups will be assessed on baseline, completion of third month after randomization (Outcome assessment), six months after randomization (first follow-up), and finally ninth months after randomization (second follow up).
  EQ-5D-5L (EuroQol, 1990) will be used to measure participant's health related quality of life across five domains i.e. mobility, self-care, usual activities, pain/discomfort and anxiety/depression on 5 levels. It also include visual analogue scale on which patient has report perceived health status on 0-100 grading.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tahir Khalily, PhD, Principal Investigator — International Islamic University, Islamabad
Locations (2):
- Pakistan (2):
  - Psychological Services Clinic, Medical Center, International Islamic University, Islamabad, Federal Capital
  - Research Office, Department of Psychology, International Islamic University Islamabad, Islamabad, Federal

IPD SHARING:
Plan to Share IPD: No